CLINICAL TRIAL: NCT00328276
Title: NMDA Enhancers in the Treatment of Schizophrenia
Brief Title: Sarcosine (N-Methylglycine) Monotherapy for Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR93-IRB-119; NHRI-EX-94-9405PI
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2006-05

CONDITIONS: Schizophrenias; Psychoses; Psychotic Disorders; Schizophrenic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Sarcosine

INTERVENTIONS:
Drug: Sarcosine

SUMMARY:
The etiology of schizophrenia remains unclear. Schizophrenia patients reveal positive symptoms, negative symptoms, and cognitive impairments. In addition to dopamine system hyperactivity, hypofunction of N-methyl-D-aspartate (NMDA) receptor plays a role in the pathophysiology of schizophrenia. Consequently, enhancing NMDA receptor neurotransmission has been considered as a novel treatment approach. To date, there have been several trials on NMDA enhancers reported. For example, sarcosine (N-methylglycine, a glycine transporter I inhibitor) showed therapeutic effects not only in chronically stable patients but also in acutely exacerbated ones when added-on to antipsychotics. In addition, sarcosine yields excellent safety profiles, in comparison to current antipsychotics.

It remains unclear whether NMDA enhancers, such as sarcosine, can serve as monotherapy for schizophrenia. The aims of this project are to examine the efficacy and safety of sarcosine monotherapy for acutely-ill schizophrenic patients, and to compare the effects of 2 grams/day, effective dose, with 1 gram/day, ineffective lower dose.

DETAILED DESCRIPTION:
In the study, 20 schizophrenic patients are recruited into the 6-week trial and randomly assigned into the two groups (1 g/d and 2 g/d) with a double-blind manner. Clinical manifestation (Positive and Negative Syndrome Scale; Scale for the Assessment of Negative Symptoms), side effects and quality of life are evaluated every two weeks during the trial. The efficacies of two groups are compared, and the characteristics of better responders are analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the criteria of schizophrenia according to the Diagnostic and Statistic Manual, fourth edition (DSM-IV).
* Free from antipsychotics for at least 7 days before enrollment.
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* Meet DSM-IV criteria of major mood disorder, current substance dependence or mental retardation
* History of epilepsy, head trauma or CNS diseases
* Major, untreated medical diseases
* Pregnancy or lactation
* Receiving psychotropic agents or depot within three months prior to study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-12; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-yuan Lane, MD,PhD, Principal Investigator — Dept. of Psychiatry, China Medical University Hospital, Taichung, Taiwan; Guochuan E. Tsai, MD,PhD, Study Director — Department of Psychiatry, Harbor-UCLA Medical Center, Torrance, California
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Lane HY, Chang YC, Liu YC, Chiu CC, Tsai GE. Sarcosine or D-serine add-on treatment for acute exacerbation of schizophrenia: a randomized, double-blind, placebo-controlled study. Arch Gen Psychiatry. 2005 Nov;62(11):1196-204. doi: 10.1001/archpsyc.62.11.1196. PMID 16275807
- [Derived] Lane HY, Liu YC, Huang CL, Chang YC, Liau CH, Perng CH, Tsai GE. Sarcosine (N-methylglycine) treatment for acute schizophrenia: a randomized, double-blind study. Biol Psychiatry. 2008 Jan 1;63(1):9-12. doi: 10.1016/j.biopsych.2007.04.038. Epub 2007 Jul 20. PMID 17659263